CLINICAL TRIAL: NCT02569190
Title: Effect of Robot-assisted Gait Training on Brain Reorganization in Hemiplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Health Service Medical Center, Seoul, Korea (Other)
Responsible Party: Principal Investigator, Dae Hyun, Medical Doctor, Veterans Health Service Medical Center, Seoul, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-05-008-002
Record Dates: First submitted 2015-09-18; First posted 2015-10-06 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Walkbot (Experimental): Receive conventional physical therapy (session I for 30 min/day) with Walkbot training 3 days a week for 8 weeks, 20 session in all.
  Interventions: Device: Walkbot

INTERVENTIONS:
Device: Walkbot — Robot assisted gait training

SUMMARY:
Purpose: To evaluate the effect of robotic gait therapy for brain reorganization in hemiplegia patients.

DETAILED DESCRIPTION:
This study designed an interventional pre-post compared clinical study. The subjects received conventional physical therapy with Walkbot training (3 sessions per week for 7 weeks, 20 session). Before and after intervention all subjects evaluated using diffusion tensor imaging and clinical outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* First stroke attack
* Within 3 months after stroke onset
* Supratentorial stroke
* Unilateral stroke

Exclusion Criteria:

* Bilateral stroke
* infratentorial stroke
* Cognitive disabilities or serious psychiatric illness.
* Difficulty in walking due to orthopedic problems.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline fraction anisotropy of corticoreticular tract in Diffusion tensor imaging 8 weeks after the first day of intervention | at the first day of intervention and 8 weeks after the first day

SECONDARY OUTCOMES:
Functional ambulation category | at the first day of intervention, 4 weeks, 8 weeks and 12 weeks after the first day
  The functional ambulation category was designed to examine the levels of assistance required during a 15m walk. Six categories are included in the functional ambulation category: 0 (non-ambulatory), 1 (needs continuous support from one person), 2 (needs intermittent support from one person), 3 (needs only verbal supervision), 4 (help is required on stairs and uneven surfaces), and 5 (can walk independently anywhere).
Fugl-meyer assessment | at the first day of intervention, 4 weeks, 8 weeks and 12 weeks after the first day
Medical research council | at the first day of intervention, 4 weeks, 8 weeks and 12 weeks after the first day
  The medical research council was designed to examine the muscle strength. Six categories are included in the medical research council: 5 (muscle contracts normally against full resistance), 4 (muscle strength is reduced but muscle contraction can still move joint against resistance), 3 (muscle strength is further reduced such that the joint can be moved only against gravity with the examiner's resistance completely removed. As an example, the elbow can be moved from full extension to full flexion starting with the arm hanging down at the side), 2 (muscle can move only if the resistance of gravity is removed. As an example, the elbow can be fully flexed only if the arm is maintained in a horizontal plane), 1 (only a trace or flicker of movement is seen or felt in the muscle or fasciculations are observed in the muscle) and 0 (no movement is observed)
Trunk control test | at the first day of intervention, 4 weeks, 8 weeks and 12 weeks after the first day

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Kim, Master, Principal Investigator — Veterans hospital, Seoul, Republic of Korea
Locations (1):
- Veterans Health Service Medical Center, Seoul, Gangdong-gu, South Korea